CLINICAL TRIAL: NCT00362895
Title: A Double-Masked, Parallel-Group, Randomized, Single-Dose Bioequivalence Study of Tobradex AF Suspension and TOBRADEX Ophthalmic Suspension
Brief Title: A Bioequivalence Study of Tobradex AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-23
Record Dates: First submitted 2006-08-09; First posted 2006-08-15 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Tobramycin; Dexamethasone; Tobramycin, Dexamethasone Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Tobradex AF (Experimental)
  Interventions: Drug: Tobramycin 0.3% / Dexamethasone 0.033% ophthalmic suspension
- TOBRADEX (Active Comparator)
  Interventions: Drug: Tobramycin 0.3% / Dexamethasone 0.1% ophthalmic suspension (TOBRADEX)

INTERVENTIONS:
Drug: Tobramycin 0.3% / Dexamethasone 0.033% ophthalmic suspension — One drop in the study eye, single dose
  Arms: Tobradex AF
Drug: Tobramycin 0.3% / Dexamethasone 0.1% ophthalmic suspension (TOBRADEX) — One drop in the study eye, single dose
  Other Names: TOBRADEX®
  Arms: TOBRADEX

SUMMARY:
The purpose of the study is to determine the amount of study medication that moves from the front of the eye into the fluid at the front of the inside of the eye.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Under 18
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 995 (Actual)
Dates: Start 2006-04; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Concentration of dexamethasone in aqueous humor following a single topical ocular administration

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon for Trial Location(s), Fort Worth, Texas, United States